CLINICAL TRIAL: NCT04656340
Title: Enhancing the Success of Functional Restoration Using Integrative Pain Therapies: a Comparative Effectiveness Analysis of Active Duty Service Members With Chronic Pain
Brief Title: Complementary and Integrative Pain Therapies and Functional Restoration (IMPPPORT) Trial)
Acronym: IMPPPORT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Madigan Army Medical Center (U.S. Federal Agency)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency); University of Washington (Other); National Institute of Nursing Research (NINR) (NIH); Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Responsible Party: Principal Investigator, Diane Flynn, Principal Investigator, Madigan Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 215050; DM140424 (Other Grant/Funding Number: US Army Medical Research and Materiel Command); K24NR015340 (NIH)
Record Dates: First submitted 2020-11-18; First posted 2020-12-07 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard rehabilitative care (SC) (Active Comparator): Twice weekly physical therapy, occupational therapy and pain psychoeducation
  Interventions: Other: non-medication, non-interventional therapies
- Complementary and Integrative Health (CIH) therapies in addition to Standard rehabilitate care (SC) (Experimental): Twice weekly chiropractic, acupuncture, yoga and foam roller instruction, in addition to SC
  Interventions: Other: non-medication, non-interventional therapies

INTERVENTIONS:
Other: non-medication, non-interventional therapies — non-medication, non-interventional therapies
  Other Names: Standard rehabilitative therapies (SC) and Complementary and Integrative Health (CIH) therapies

SUMMARY:
This study aims to evaluate the benefit of a complementary and integrative health (CIH) pain management program when added to standard rehabilitative care (SC) compared to SC alone prior to an intensive functional restoration (FR) program in a population of active duty service members. In addition the study aims to identify factors that predict improvement in pain impact following treatment, and to determine the proportion of participants who experience clinically meaningful response.

SC included physical and occupational therapy. CIH included chiropractic, acupuncture, yoga and foam roller instruction. Both treatment groups also received education about pain psychology.

Participants were randomly assigned to a 3-week course of either SC alone or CIH combined with SC prior to a 3-week course of FR. Outcomes were collected at baseline, at end of stage 1, and post-FR. Outcomes included patient-reported and provider-determined measures.

ELIGIBILITY:
Inclusion Criteria:

* Significant functional impairment due to pain, requiring modification of military duties.
* Physically able to participate in up to four hours of physical activity (strength, flexibility, endurance training) per day:

  1. Can stand up from and sit down on floor independently
  2. Can walk on treadmill for at least 6 minutes at 2.5 mile/hour pace or faster.
  3. Able to complete at least 2 of the following:

     1. Lift 20 lbs from floor to knuckle height
     2. Lift 20 lbs from floor to shoulder height
     3. Carry 20lbs at least 40 feet.
* Inadequate response to previous less intensive treatment
* Expresses motivation to take active role in regaining function

Exclusion Criteria:

* Major surgeries within past 6 months or planned within next 6 months
* Unstable psychological disorders
* Active substance use disorder
* High dose opioids of >120 milligrams of morphine equivalent doses (MED)/day

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2015-12-09 (Actual); Primary Completion 2019-04-02 (Actual); Study Completion 2019-04-02 (Actual)

PRIMARY OUTCOMES:
Change in National Institutes of Health (NIH) Research Task Force (RTF) Impact Score - baseline to end of stage 1 treatment | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. End of stage 1 measures collected between </=2 treatment days before end of stage 1 through 4 treatment days after end of stage 1.
  The RTF Impact score is was computed by adding the following three scores: 1) average pain intensity (range 0=no pain - 10=worst pain) from the Defense and Veterans Pain Rating Scale (DVPRS); 2) the NIH Patient Reported Outcome Measures Information System (PROMIS) pain interference score (range 4-20 with higher scores indicating worse status; 3) the REVERSE of the PROMIS physical function scores (range 4-20 with higher score indicating better status and higher score on reverse scale indicating worse status). The range of RTF impact score is 8 (best) -50 (worst). Change in Impact Score is computed by subtracting baseline Impact Score from the score at the time of reassessment. Improvement is indicated by change scores with negative values.
Change in National Institutes of Health (NIH) Research Task Force (RTF) Impact Score - baseline to end of stage 2 treatment | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. End of Stage 2 measures collected between </=2 treatment days before end of stage 2 through 30 days after end of stage 2.
  The RTF Impact score is was computed by adding the following three scores: 1) average pain intensity (range 0=no pain - 10=worst pain) from the Defense and Veterans Pain Rating Scale (DVPRS); 2) the NIH Patient Reported Outcome Measures Information System (PROMIS) pain interference score (range 4-20 with higher scores indicating worse status; 3) the REVERSE of the PROMIS physical function scores (range 4-20 with higher score indicating better status and higher score on reverse scale indicating worse status). The range of RTF impact score is 8 (best) -50 (worst). Change in RTF Impact Score from baseline to end of stage 2

SECONDARY OUTCOMES:
Change in National Institutes of Health (NIH) Research Task Force (RTF) Impact Score - short-term follow-up | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. Short-term follow-up measures collected between 1 month through <5 months after end of stage 2.
  The RTF Impact score is was computed by adding the following three scores: 1) average pain intensity (range 0=no pain - 10=worst pain) from the Defense and Veterans Pain Rating Scale (DVPRS); 2) the NIH Patient Reported Outcome Measures Information System (PROMIS) pain interference score (range 4-20 with higher scores indicating worse status; 3) the REVERSE of the PROMIS physical function scores (range 4-20 with higher score indicating better status and higher score on reverse scale indicating worse status). The range of RTF impact score is 8 (best) -50 (worst). Change in RTF Impact Score from baseline to short-term post-treatment follow-up.
Change in National Institutes of Health (NIH) Research Task Force (RTF) Impact Score - intermediate-term follow-up | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. Intermediate-term follow-up measures collected between >6 month through <9 months after end of stage 2.
  The RTF Impact score is was computed by adding the following three scores: 1) average pain intensity (range 0=no pain - 10=worst pain) from the Defense and Veterans Pain Rating Scale (DVPRS); 2) the NIH Patient Reported Outcome Measures Information System (PROMIS) pain interference score (range 4-20 with higher scores indicating worse status; 3) the REVERSE of the PROMIS physical function scores (range 4-20 with higher score indicating better status and higher score on reverse scale indicating worse status). The range of RTF impact score is 8 (best) -50 (worst). Change in RTF Impact Score from baseline to intermediate-term post-treatment follow-up.
Battery of functional performance measures - Change in walking tolerance from baseline to end of stage 1 | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. End of stage 1 measures collected between </=2 treatment days before end of stage 1 through 4 treatment days after end of stage 1.
  Walking tolerance on a treadmill using the modified Naughton treadmill protocol. Measured in minutes completed. Higher number of minutes indicates better status. Test terminates when pain intensity increases from level at start of treadmill testing. Change score is computed by subtracting the baseline number of minutes completed from the number of minutes completed at the time of reassessment. Improvement is indicated by change scores with positive values.
Battery of functional performance measures - Change in walking tolerance from baseline to end of stage 2 | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. End of Stage 2 measures collected between </=2 treatment days before end of stage 2 through 30 days after end of stage 2.
  Walking tolerance on a treadmill using the modified Naughton treadmill protocol. Measured in minutes completed. Higher number of minutes indicates better status. Test terminates when pain intensity increases from level at start of treadmill testing. Change score is computed by subtracting the baseline number of minutes completed from the number of minutes completed at the time of reassessment. Improvement is indicated by change scores with positive values.
Battery of functional performance measures - Change in walking tolerance from baseline to short-term post-treatment follow-up. | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. Short-term follow-up measures collected between 1 month through <5 months after end of stage 2.
  Walking tolerance on a treadmill using the modified Naughton treadmill protocol. Measured in minutes completed. Higher number of minutes indicates better status. Test terminates when pain intensity increases from level at start of treadmill testing. Change score is computed by subtracting the baseline number of minutes completed from the number of minutes completed at the time of reassessment. Improvement is indicated by change scores with positive values.
Battery of functional performance measures - Change in walking tolerance from baseline to intermediate-term post-treatment follow-up | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. Intermediate-term follow-up measures collected between >6 month through <9 months after end of stage 2.
  Walking tolerance on a treadmill using the modified Naughton treadmill protocol. Measured in minutes completed. Higher number of minutes indicates better status. Test terminates when pain intensity increases from level at start of treadmill testing. Change score is computed by subtracting the baseline number of minutes completed from the number of minutes completed at the time of reassessment. Improvement is indicated by change scores with positive values.
Battery of functional performance measures - Change in floor-to-waist lifting tolerance from baseline to end of Stage 1. Improvement is indicated by change scores with positive values. | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. End of stage 1 measures collected between </=2 treatment days before end of stage 1 through 4 treatment days after end of stage 1.
  Measures how much weight in pounds study subject can comfortably lift from floor to waist height. Higher number of lbs lifted indicates better status. Test terminates when pain intensity increases from start of lift test. Change score is measured in pounds and is computed by subtracting the baseline number of pounds lifted from the number of pounds lifted at time of reassessment. Improvement is indicated by change scores with positive values.
Battery of functional performance measures - Change in floor-to-waist lifting tolerance from baseline to end of Stage 2 | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. End of Stage 2 measures collected between </=2 treatment days before end of stage 2 through 30 days after end of stage 2.
  Measures how much weight in pounds study subject can comfortably lift from floor to waist height. Higher number of lbs lifted indicates better status. Test terminates when pain intensity increases from start of lift test. Change score is measured in pounds and is computed by subtracting the baseline number of pounds lifted from the number of pounds lifted at time of reassessment. Improvement is indicated by change scores with positive values.
Battery of functional performance measures - Change in floor-to-waist lifting tolerance from baseline to end of short-term post-treatment follow-up | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. Short-term follow-up measures collected between 1 month through <5 months after end of stage 2.
  Measures how much weight in pounds study subject can comfortably lift from floor to waist height. Higher number of lbs lifted indicates better status. Test terminates when pain intensity increases from start of lift test. Change score is measured in pounds and is computed by subtracting the baseline number of pounds lifted from the number of pounds lifted at time of reassessment. Improvement is indicated by change scores with positive values.
Battery of functional performance measures - Change in floor-to-waist lifting tolerance from baseline to end of intermediate-term post-treatment follow-up | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. Intermediate-term follow-up measures collected between >6 month through <9 months after end of stage 2.
  Measures how much weight in pounds study subject can comfortably lift from floor to waist height. Higher number of lbs lifted indicates better status. Test terminates when pain intensity increases from start of lift test. Change score is measured in pounds and is computed by subtracting the baseline number of pounds lifted from the number of pounds lifted at time of reassessment. Improvement is indicated by change scores with positive values.
Battery of functional performance measures - Change in waist-shoulder lifting tolerance from baseline to end of stage-1. | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. End of stage 1 measures collected between </=2 treatment days before end of stage 1 through 4 treatment days after end of stage 1.
  Measures how much weight in pounds study subject can comfortably lift from waist to shoulder height. Higher number of lbs lifted indicates better status. Test terminates when pain intensity increases from start of lift test. Change score is measured in pounds and is computed by subtracting the baseline number of pounds lifted from the number of pounds lifted at time of reassessment. Improvement is indicated by change scores with positive values.
Battery of functional performance measures - Change in waist-shoulder lifting tolerance from baseline to end of stage-2. | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. End of Stage 2 measures collected between </=2 treatment days before end of stage 2 through 30 days after end of stage 2.
  Measures how much weight in pounds study subject can comfortably lift from waist to shoulder height. Higher number of lbs lifted indicates better status. Test terminates when pain intensity increases from start of lift test. Change score is measured in pounds and is computed by subtracting the baseline number of pounds lifted from the number of pounds lifted at time of reassessment. Improvement is indicated by change scores with positive values.
Battery of functional performance measures - Change in waist-shoulder lifting tolerance from baseline to short-term post-treatment follow-up. | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. Short-term follow-up measures collected between 1 month through <5 months after end of stage 2.
  Measures how much weight in pounds study subject can comfortably lift from waist to shoulder height. Higher number of lbs lifted indicates better status. Test terminates when pain intensity increases from start of lift test. Change score is measured in pounds and is computed by subtracting the baseline number of pounds lifted from the number of pounds lifted at time of reassessment. Improvement is indicated by change scores with positive values.
Battery of functional performance measures - Change in waist-shoulder lifting tolerance from baseline to intermediate-term post-treatment follow-up. | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. Intermediate-term follow-up measures collected between >6 month through <9 months after end of stage 2.
  Measures how much weight in pounds study subject can comfortably lift from waist to shoulder height. Higher number of lbs lifted indicates better status. Test terminates when pain intensity increases from start of lift test. Change score is measured in pounds and is computed by subtracting the baseline number of pounds lifted from the number of pounds lifted at time of reassessment. Improvement is indicated by change scores with positive values.
Battery of functional performance measures - Change in 40-foot carry tolerance from baseline to end of stage 1 | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. End of stage 1 measures collected between </=2 treatment days before end of stage 1 through 4 treatment days after end of stage 1.
  Measures how much weight in pounds study subject can carry a distance of 40-feet. Higher number of lbs carried indicates better status. Test terminates when pain intensity increases from start of carry test. Change score is measured in pounds and is computed by subtracting the baseline number of pounds carried from the number of pounds lifted at time of reassessment. Improvement is indicated by change scores with positive values.
Battery of functional performance measures - Change in 40-foot carry tolerance from baseline to end of stage 2. | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. End of Stage 2 measures collected between </=2 treatment days before end of stage 2 through 30 days after end of stage 2.
  Measures how much weight in pounds study subject can carry a distance of 40-feet. Higher number of lbs carried indicates better status. Test terminates when pain intensity increases from start of carry test. Change score is measured in pounds and is computed by subtracting the baseline number of pounds carried from the number of pounds lifted at time of reassessment. Improvement is indicated by change scores with positive values.
Battery of functional performance measures - Change in 40-foot carry tolerance from baseline to short-term post-treatment follow-up. | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. Short-term follow-up measures collected between 1 month through <5 months after end of stage 2.
  Measures how much weight in pounds study subject can carry a distance of 40-feet. Higher number of lbs carried indicates better status. Test terminates when pain intensity increases from start of carry test. Change score is measured in pounds and is computed by subtracting the baseline number of pounds carried from the number of pounds lifted at time of reassessment. Improvement is indicated by change scores with positive values.
Battery of functional performance measures - Change in 40-foot carry tolerance from baseline to intermediate-term post-treatment follow-up. | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. Intermediate-term follow-up measures collected between >6 month through <9 months after end of stage 2.
  Measures how much weight in pounds study subject can carry a distance of 40-feet. Higher number of lbs carried indicates better status. Test terminates when pain intensity increases from start of carry test. Change score is measured in pounds and is computed by subtracting the baseline number of pounds carried from the number of pounds lifted at time of reassessment. Improvement is indicated by change scores with positive values.
Change in NIH Patient Reported Outcome Measures Information System (PROMIS) Depression - baseline to end of stage 1 | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. End of stage 1 measures collected between </=2 treatment days before end of stage 1 through 4 treatment days after end of stage 1.
  PROMIS Depression reported in T-score, range 0-100, with 50 corresponding to the mean score and higher scores indicate worse depression. Change score is computed by subtracting baseline Depression T-score from T-score at time of reassessment. Improvement is indicated by change scores with negative values.
Change in NIH Patient Reported Outcome Measures Information System (PROMIS) Depression - baseline to end of stage 2 | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. End of Stage 2 measures collected between </=2 treatment days before end of stage 2 through 30 days after end of stage 2.
  PROMIS Depression reported in T-score, range 0-100, with 50 corresponding to the mean score and higher scores indicate worse depression. Change score is computed by subtracting baseline Depression T-score from T-score at time of reassessment. Improvement is indicated by change scores with negative values.
Change in NIH Patient Reported Outcome Measures Information System (PROMIS) Depression - baseline to short-term post-treatment follow-up | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. Short-term follow-up measures collected between 1 month through <5 months after end of stage 2.
  PROMIS Depression reported in T-score, range 0-100, with 50 corresponding to the mean score and higher scores indicate worse depression. Change score is computed by subtracting baseline Depression T-score from T-score at time of reassessment. Improvement is indicated by change scores with negative values.
Change in NIH Patient Reported Outcome Measures Information System (PROMIS) Depression - baseline to intermediate-term post-treatment follow-up | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. Intermediate-term follow-up measures collected between >6 month through <9 months after end of stage 2.
  PROMIS Depression reported in T-score, range 0-100, with 50 corresponding to the mean score and higher scores indicate worse depression. Change score is computed by subtracting baseline Depression T-score from T-score at time of reassessment. Improvement is indicated by change scores with negative values.
Change in NIH Patient Reported Outcome Measures Information System (PROMIS) Anxiety - baseline to end of stage 1. | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. End of stage 1 measures collected between </=2 treatment days before end of stage 1 through 4 treatment days after end of stage 1.
  PROMIS Anxiety reported in T-score, range 0-100, with 50 corresponding to the mean score and higher scores indicate worse anxiety. Change score is computed by subtracting baseline Anxiety T-score from T-score at time of reassessment. Improvement is indicated by change scores with negative values.
Change in NIH Patient Reported Outcome Measures Information System (PROMIS) Anxiety - baseline to end of stage 2. | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. End of Stage 2 measures collected between </=2 treatment days before end of stage 2 through 30 days after end of stage 2.
  PROMIS Anxiety reported in T-score, range 0-100, with 50 corresponding to the mean score and higher scores indicate worse anxiety. Change score is computed by subtracting baseline Anxiety T-score from T-score at time of reassessment. Improvement is indicated by change scores with negative values.
Change in NIH Patient Reported Outcome Measures Information System (PROMIS) Anxiety - baseline to short-term post-treatment follow-up | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. Short-term follow-up measures collected between 1 month through <5 months after end of stage 2.
  PROMIS Anxiety reported in T-score, range 0-100, with 50 corresponding to the mean score and higher scores indicate worse anxiety. Change score is computed by subtracting baseline Anxiety T-score from T-score at time of reassessment. Improvement is indicated by change scores with negative values.
Change in NIH Patient Reported Outcome Measures Information System (PROMIS) Anxiety - baseline to intermediate-term post-treatment follow-up | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. Intermediate-term follow-up measures collected between >6 month through <9 months after end of stage 2.
  PROMIS Anxiety reported in T-score, range 0-100, with 50 corresponding to the mean score and higher scores indicate worse anxiety. Change score is computed by subtracting baseline Anxiety T-score from T-score at time of reassessment. Improvement is indicated by change scores with negative values.
Change in NIH Patient Reported Outcome Measures Information System (PROMIS) Anger - baseline to end of stage 1 | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. End of stage 1 measures collected between </=2 treatment days before end of stage 1 through 4 treatment days after end of stage 1.
  PROMIS Anger reported in T-score, range 0-100, with 50 corresponding to the mean score and higher scores indicate worse anxiety. Change score is computed by subtracting baseline Anger T-score from T-score at time of reassessment. Improvement is indicated by change scores with negative values.
Change in NIH Patient Reported Outcome Measures Information System (PROMIS) Anger - baseline to intermediate-term post-treatment follow-up | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. End of Stage 2 measures collected between </=2 treatment days before end of stage 2 through 30 days after end of stage 2.
  PROMIS Anger reported in T-score, range 0-100, with 50 corresponding to the mean score and higher scores indicate worse anxiety. Change score is computed by subtracting baseline Anger T-score from T-score at time of reassessment. Improvement is indicated by change scores with negative values.
Change in NIH Patient Reported Outcome Measures Information System (PROMIS) Anger - baseline to intermediate-term post-treatment follow-up | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. Short-term follow-up measures collected between 1 month through <5 months after end of stage 2.
  PROMIS Anger reported in T-score, range 0-100, with 50 corresponding to the mean score and higher scores indicate worse anxiety. Change score is computed by subtracting baseline Anger T-score from T-score at time of reassessment. Improvement is indicated by change scores with negative values.
Change in NIH Patient Reported Outcome Measures Information System (PROMIS) Anger - baseline to intermediate-term post-treatment follow-up | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. Intermediate-term follow-up measures collected between >6 month through <9 months after end of stage 2.
  PROMIS Anger reported in T-score, range 0-100, with 50 corresponding to the mean score and higher scores indicate worse anxiety. Change score is computed by subtracting baseline Anger T-score from T-score at time of reassessment. Improvement is indicated by change scores with negative values.
Change in NIH Patient Reported Outcome Measures Information System (PROMIS) Sleep-related Impairment - baseline to end of stage 1 | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. End of stage 1 measures collected between </=2 treatment days before end of stage 1 through 4 treatment days after end of stage 1.
  PROMIS Sleep-related Impairment reported in T-score, range 0-100, with 50 corresponding to the mean score and higher scores indicate worse Sleep-related Impairment. Change score is computed by subtracting baseline Sleep-related Impairment T-score from T-score at time of reassessment. Improvement is indicated by change scores with negative values.
Change in NIH Patient Reported Outcome Measures Information System (PROMIS) Sleep-related Impairment - baseline to end of stage 2 | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. End of Stage 2 measures collected between </=2 treatment days before end of stage 2 through 30 days after end of stage 2.
  PROMIS Sleep-related Impairment reported in T-score, range 0-100, with 50 corresponding to the mean score and higher scores indicate worse Sleep-related Impairment. Change score is computed by subtracting baseline Sleep-related Impairment T-score from T-score at time of reassessment. Improvement is indicated by change scores with negative values.
Change in NIH Patient Reported Outcome Measures Information System (PROMIS) Sleep-related Impairment - baseline to short-term post-treatment follow-up | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. Short-term follow-up measures collected between 1 month through <5 months after end of stage 2.
  PROMIS Sleep-related Impairment reported in T-score, range 0-100, with 50 corresponding to the mean score and higher scores indicate worse Sleep-related Impairment. Change score is computed by subtracting baseline Sleep-related Impairment T-score from T-score at time of reassessment. Improvement is indicated by change scores with negative values.
Change in NIH Patient Reported Outcome Measures Information System (PROMIS) Sleep-related Impairment - baseline to intermediate-term post-treatment follow-up | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. Intermediate-term follow-up measures collected between >6 month through <9 months after end of stage 2.
  PROMIS Sleep-related Impairment reported in T-score, range 0-100, with 50 corresponding to the mean score and higher scores indicate worse Sleep-related Impairment. Change score is computed by subtracting baseline Sleep-related Impairment T-score from T-score at time of reassessment. Improvement is indicated by change scores with negative values.
Change in NIH Patient Reported Outcome Measures Information System (PROMIS) Physical Function - baseline to end of stage 1. | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. End of stage 1 measures collected between </=2 treatment days before end of stage 1 through 4 treatment days after end of stage 1.
  PROMIS Sleep-related Impairment reported in T-score, range 0-100, with 50 corresponding to the mean score and higher scores indicate better physical function. Change score is computed by subtracting baseline Sleep-related Impairment T-score from T-score at time of reassessment. Improvement is indicated by change scores with positive values.
Change in NIH Patient Reported Outcome Measures Information System (PROMIS) Physical Function - baseline to end of stage 2. | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. End of Stage 2 measures collected between </=2 treatment days before end of stage 2 through 30 days after end of stage 2.
  PROMIS Sleep-related Impairment reported in T-score, range 0-100, with 50 corresponding to the mean score and higher scores indicate better physical function. Change score is computed by subtracting baseline Sleep-related Impairment T-score from T-score at time of reassessment. Improvement is indicated by change scores with positive values.
Change in NIH Patient Reported Outcome Measures Information System (PROMIS) Physical Function - baseline to short-term post-treatment follow-up | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. Short-term follow-up measures collected between 1 month through <5 months after end of stage 2.
  PROMIS Sleep-related Impairment reported in T-score, range 0-100, with 50 corresponding to the mean score and higher scores indicate better physical function. Change score is computed by subtracting baseline Sleep-related Impairment T-score from T-score at time of reassessment. Improvement is indicated by change scores with positive values.
Change in NIH Patient Reported Outcome Measures Information System (PROMIS) Physical Function - baseline to intermediate-term post-treatment follow-up | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. Intermediate-term follow-up measures collected between >6 month through <9 months after end of stage 2.
  PROMIS Sleep-related Impairment reported in T-score, range 0-100, with 50 corresponding to the mean score and higher scores indicate better physical function. Change score is computed by subtracting baseline Sleep-related Impairment T-score from T-score at time of reassessment. Improvement is indicated by change scores with positive values.
Change in NIH Patient Reported Outcome Measures Information System (PROMIS) Satisfaction with Social Roles - baseline to end of stage 1. | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. End of stage 1 measures collected between </=2 treatment days before end of stage 1 through 4 treatment days after end of stage 1.
  PROMIS Satisfaction with Social Roles reported in T-score, range 0-100, with 50 corresponding to the mean score and higher scores indicate better satisfaction with social roles. Change score is computed by subtracting baseline Sleep-related Impairment T-score from T-score at time of reassessment. Improvement is indicated by change scores with positive values.
Change in NIH Patient Reported Outcome Measures Information System (PROMIS) Satisfaction with Social Roles - baseline to end of stage 2 | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. End of Stage 2 measures collected between </=2 treatment days before end of stage 2 through 30 days after end of stage 2.
  PROMIS Satisfaction with Social Roles reported in T-score, range 0-100, with 50 corresponding to the mean score and higher scores indicate better satisfaction with social roles. Change score is computed by subtracting baseline Sleep-related Impairment T-score from T-score at time of reassessment. Improvement is indicated by change scores with positive values.
Change in NIH Patient Reported Outcome Measures Information System (PROMIS) Satisfaction with Social Roles - baseline to short-term post-treatment follow-up | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. Short-term follow-up measures collected between 1 month through <5 months after end of stage 2.
  PROMIS Satisfaction with Social Roles reported in T-score, range 0-100, with 50 corresponding to the mean score and higher scores indicate better satisfaction with social roles. Change score is computed by subtracting baseline Sleep-related Impairment T-score from T-score at time of reassessment. Improvement is indicated by change scores with positive values.
Change in NIH Patient Reported Outcome Measures Information System (PROMIS) Satisfaction with Social Roles - baseline to intermediate-term post-treatment follow-up | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. Intermediate-term follow-up measures collected between >6 month through <9 months after end of stage 2.
  PROMIS Satisfaction with Social Roles reported in T-score, range 0-100, with 50 corresponding to the mean score and higher scores indicate better satisfaction with social roles. Change score is computed by subtracting baseline Sleep-related Impairment T-score from T-score at time of reassessment. Improvement is indicated by change scores with positive values.
Change in Pain Catastrophizing Score (PCS), baseline to end of stage 1 | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. End of stage 1 measures collected between </=2 treatment days before end of stage 1 through 4 treatment days after end of stage 1.
  PCS is a 13-item questionnaire with a score range 0-52 with higher scores indicating worse status. Change score is computed by subtracting baseline PCS from PCS at time of reassessment. Improvement is indicated by change scores with negative values.
Change in Pain Catastrophizing Score (PCS), baseline to end of stage 2 | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. End of Stage 2 measures collected between </=2 treatment days before end of stage 2 through 30 days after end of stage 2.
  PCS is a 13-item questionnaire with a score range 0-52 with higher scores indicating worse status. Change score is computed by subtracting baseline PCS from PCS at time of reassessment. Improvement is indicated by change scores with negative values.
Change in Pain Catastrophizing Score (PCS), baseline to short-term follow-up | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. Short-term follow-up measures collected between 1 month through <5 months after end of stage 2.
  PCS is a 13-item questionnaire with a score range 0-52 with higher scores indicating worse status. Change score is computed by subtracting baseline PCS from PCS at time of reassessment. Improvement is indicated by change scores with negative values.
Change in Pain Catastrophizing Score (PCS), baseline to intermediate-term follow-up | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. Intermediate-term follow-up measures collected between >6 month through <9 months after end of stage 2.
  PCS is a 13-item questionnaire with a score range 0-52 with higher scores indicating worse status. Change score is computed by subtracting baseline PCS from PCS at time of reassessment. Improvement is indicated by change scores with negative values.
Change in Chronic Pain Acceptance Questionnaire-8 (CPAQ-8), baseline to end of stage 1 | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. End of stage 1 measures collected between </=2 treatment days before end of stage 1 through 4 treatment days after end of stage 1.
  CPAQ-8 is an 8-item questionnaire with a score range 0-48 with higher scores indicating better status. Change score is computed by subtracting baseline CPAQ-8 score from score at time of reassessment. Improvement is indicated by change scores with positive values.
Change in Chronic Pain Acceptance Questionnaire-8 (CPAQ-8), baseline to end of stage 2 | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. End of Stage 2 measures collected between </=2 treatment days before end of stage 2 through 30 days after end of stage 2.
  CPAQ-8 is an 8-item questionnaire with a score range 0-48 with higher scores indicating better status. Change score is computed by subtracting baseline CPAQ-8 score from score at time of reassessment. Improvement is indicated by change scores with positive values.
Change in Chronic Pain Acceptance Questionnaire-8 (CPAQ-8), baseline to short-term follow-up | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. Short-term follow-up measures collected between 1 month through <5 months after end of stage 2.
  CPAQ-8 is an 8-item questionnaire with a score range 0-48 with higher scores indicating better status. Change score is computed by subtracting baseline CPAQ-8 score from score at time of reassessment. Improvement is indicated by change scores with positive values.
Change in Chronic Pain Acceptance Questionnaire-8 (CPAQ-8), baseline to intermediate-term follow-up | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. Intermediate-term follow-up measures collected between >6 month through <9 months after end of stage 2.
  CPAQ-8 is an 8-item questionnaire with a score range 0-48 with higher scores indicating better status. Change score is computed by subtracting baseline CPAQ-8 score from score at time of reassessment. Improvement is indicated by change scores with positive values.
Change in Pain Self-Efficacy Questionnaire (PSEQ), baseline to end of stage 1 | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. End of stage 1 measures collected between </=2 treatment days before end of stage 1 through 4 treatment days after end of stage 1.
  PSEQ is a 10-item questionnaire with a score range 0-60 with higher scores indicating better status. Change score is computed by subtracting baseline PSEQ score from score at time of reassessment. Improvement is indicated by change scores with positive values.
Change in Pain Self-Efficacy Questionnaire (PSEQ), baseline to end of stage 2 | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. End of Stage 2 measures collected between </=2 treatment days before end of stage 2 through 30 days after end of stage 2.
  PSEQ is a 10-item questionnaire with a score range 0-60 with higher scores indicating better status. Change score is computed by subtracting baseline PSEQ score from score at time of reassessment. Improvement is indicated by change scores with positive values.
Change in Pain Self-Efficacy Questionnaire (PSEQ), baseline to short-term follow-up | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. Short-term follow-up measures collected between 1 month through <5 months after end of stage 2.
  PSEQ is a 10-item questionnaire with a score range 0-60 with higher scores indicating better status. Change score is computed by subtracting baseline PSEQ score from score at time of reassessment. Improvement is indicated by change scores with positive values.
Change in Pain Self-Efficacy Questionnaire (PSEQ), baseline to intermediate-term follow-up | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. Intermediate-term follow-up measures collected between >6 month through <9 months after end of stage 2.
  PSEQ is a 10-item questionnaire with a score range 0-60 with higher scores indicating better status. Change score is computed by subtracting baseline PSEQ score from score at time of reassessment. Improvement is indicated by change scores with positive values.
Change in Patient Activation Measure (PAM), baseline to end of stage 1 | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. End of stage 1 measures collected between </=2 treatment days before end of stage 1 through 4 treatment days after end of stage 1.
  PAM a 10-item questionnaire with a score range 10-40 with higher scores indicating better status. Change score is computed by subtracting baseline PAM score from score at time of reassessment. Improvement is indicated by change scores with positive values.
Change in Patient Activation Measure (PAM), baseline to end of stage 2 | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. End of Stage 2 measures collected between </=2 treatment days before end of stage 2 through 30 days after end of stage 2.
  PAM a 10-item questionnaire with a score range 10-40 with higher scores indicating better status. Change score is computed by subtracting baseline PAM score from score at time of reassessment. Improvement is indicated by change scores with positive values.
Change in Patient Activation Measure (PAM), baseline to short-term follow-up | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. Short-term follow-up measures collected between 1 month through <5 months after end of stage 2.
  PAM a 10-item questionnaire with a score range 10-40 with higher scores indicating better status. Change score is computed by subtracting baseline PAM score from score at time of reassessment. Improvement is indicated by change scores with positive values.
Change in Patient Activation Measure (PAM), baseline to intermediate-term follow-up | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. Intermediate-term follow-up measures collected between >6 month through <9 months after end of stage 2.
  PAM a 10-item questionnaire with a score range 10-40 with higher scores indicating better status. Change score is computed by subtracting baseline PAM score from score at time of reassessment. Improvement is indicated by change scores with positive values.
Change in Tampa Kinesiophobia Score-11 (TSK-11), baseline to end of stage 1 | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. End of stage 1 measures collected between </=2 treatment days before end of stage 1 through 4 treatment days after end of stage 1.
  TSK-11 an 11-item questionnaire with a score range 11-44 with higher scores indicating worse status. Change score is computed by subtracting baseline TSK-11 score from score at time of reassessment. Improvement is indicated by change scores with negative values.
Change in Tampa Kinesiophobia Score-11 (TSK-11), baseline to end of stage 2 | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. End of Stage 2 measures collected between </=2 treatment days before end of stage 2 through 30 days after end of stage 2.
  TSK-11 an 11-item questionnaire with a score range 11-44 with higher scores indicating worse status. Change score is computed by subtracting baseline TSK-11 score from score at time of reassessment. Improvement is indicated by change scores with negative values.
Change in Tampa Kinesiophobia Score-11 (TSK-11), baseline to short-term follow-up | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. Short-term follow-up measures collected between 1 month through <5 months after end of stage 2.
  TSK-11 an 11-item questionnaire with a score range 11-44 with higher scores indicating worse status. Change score is computed by subtracting baseline TSK-11 score from score at time of reassessment. Improvement is indicated by change scores with negative values.
Change in Tampa Kinesiophobia Score-11 (TSK-11), baseline to intermediate-term follow-up | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. Intermediate-term follow-up measures collected between >6 month through <9 months after end of stage 2.
  TSK-11 an 11-item questionnaire with a score range 11-44 with higher scores indicating worse status. Change score is computed by subtracting baseline TSK-11 score from score at time of reassessment. Improvement is indicated by change scores with negative values.
Change in Roland-Morris Disability Questionnaire (RMDQ), baseline to end of stage 1 | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. End of stage 1 measures collected between </=2 treatment days before end of stage 1 through 4 treatment days after end of stage 1.
  RMDQ a 24-item questionnaire with a score range 0-24 with higher scores indicating worse status. Change score is computed by subtracting baseline RMDQ score from score at time of reassessment. Improvement is indicated by change scores with negative values.
Change in Roland-Morris Disability Questionnaire (RMDQ), baseline to of stage 2 | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. End of Stage 2 measures collected between </=2 treatment days before end of stage 2 through 30 days after end of stage 2.
  RMDQ a 24-item questionnaire with a score range 0-24 with higher scores indicating worse status. Change score is computed by subtracting baseline RMDQ score from score at time of reassessment. Improvement is indicated by change scores with negative values.
Change in Roland-Morris Disability Questionnaire (RMDQ), baseline to short-term follow-up | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. Short-term follow-up measures collected between 1 month through <5 months after end of stage 2.
  RMDQ a 24-item questionnaire with a score range 0-24 with higher scores indicating worse status. Change score is computed by subtracting baseline RMDQ score from score at time of reassessment. Improvement is indicated by change scores with negative values.
Change in Roland-Morris Disability Questionnaire (RMDQ), baseline to intermediate-term follow-up | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. Intermediate-term follow-up measures collected between >6 month through <9 months after end of stage 2.
  RMDQ a 24-item questionnaire with a score range 0-24 with higher scores indicating worse status. Change score is computed by subtracting baseline RMDQ score from score at time of reassessment. Improvement is indicated by change scores with negative values.
Patient Global Impression of Change (PGIC) at end of Stage 2 | End of Stage 2 timeline parameters as stated for outcomes 2
  PGIC is a one-item questionnaire that determines the study subjects' assessment on their level of improvement or worsening since the start of treatment. Responses are on a likert scale from very much improved; much improved; minimally improved; no change; minimally worse; much worse; very much worse
Change in Pyramid Measure, baseline to end of stage 1 | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. End of stage 1 measures collected between </=2 treatment days before end of stage 1 through 4 treatment days after end of stage 1.
  7-to-1 Pyramid Test is a functional performance test that measures the number of repetitions a person can do of sets of pushups, back extensions, rowers, squats, dips, and burpees. The total score is the total repetitions completed within 5 minutes. The minimum score is zero repetitions; there is no maximum number of repetitions. A higher number of repetitions indicates better functional status. Change score is computed by subtracting baseline number or repetitions from score at time of reassessment. Improvement is indicated by change scores with positive values.
Change in Pyramid Measure, baseline to end of stage 2 | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. End of Stage 2 measures collected between </=2 treatment days before end of stage 2 through 30 days after end of stage 2.
  7-to-1 Pyramid Test is a functional performance test that measures the number of repetitions a person can do of sets of pushups, back extensions, rowers, squats, dips, and burpees. The total score is the total repetitions completed within 5 minutes. The minimum score is zero repetitions; there is no maximum number of repetitions. A higher number of repetitions indicates better functional status. Change score is computed by subtracting baseline number or repetitions from score at time of reassessment. Improvement is indicated by change scores with positive values.
Change in Pyramid Measure, baseline to short-term follow-up | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. Short-term follow-up measures collected between 1 month through <5 months after end of stage 2.
  7-to-1 Pyramid Test is a functional performance test that measures the number of repetitions a person can do of sets of pushups, back extensions, rowers, squats, dips, and burpees. The total score is the total repetitions completed within 5 minutes. The minimum score is zero repetitions; there is no maximum number of repetitions. A higher number of repetitions indicates better functional status. Change score is computed by subtracting baseline number or repetitions from score at time of reassessment. Improvement is indicated by change scores with positive values.
Change in Pyramid Measure, baseline to intermediate-term follow-up | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. Intermediate-term follow-up measures collected between >6 month through <9 months after end of stage 2.
  7-to-1 Pyramid Test is a functional performance test that measures the number of repetitions a person can do of sets of pushups, back extensions, rowers, squats, dips, and burpees. The total score is the total repetitions completed within 5 minutes. The minimum score is zero repetitions; there is no maximum number of repetitions. A higher number of repetitions indicates better functional status. Change score is computed by subtracting baseline number or repetitions from score at time of reassessment. Improvement is indicated by change scores with positive values.
Change in NIH Patient Reported Outcome Measures Information System (PROMIS) Fatigue, baseline to end of stage 1 | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. End of stage 1 measures collected between </=2 treatment days before end of stage 1 through 4 treatment days after end of stage 1.
  PROMIS Fatigue reported in T-score, range 0-100, with 50 corresponding to the mean score and higher scores indicate worse fatigue. Change score is computed by subtracting baseline Fatigue T-score from T-score at time of reassessment. Improvement is indicated by change scores with negative values.
Change in NIH Patient Reported Outcome Measures Information System (PROMIS) Fatigue, baseline to end of stage 2 | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. End of Stage 2 measures collected between </=2 treatment days before end of stage 2 through 30 days after end of stage 2.
  PROMIS Fatigue reported in T-score, range 0-100, with 50 corresponding to the mean score and higher scores indicate worse fatigue. Change score is computed by subtracting baseline Fatigue T-score from T-score at time of reassessment. Improvement is indicated by change scores with negative values.
Change in NIH Patient Reported Outcome Measures Information System (PROMIS) Fatigue, baseline to end of short-term follow-up | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. Short-term follow-up measures collected between 1 month through <5 months after end of stage 2.
  PROMIS Fatigue reported in T-score, range 0-100, with 50 corresponding to the mean score and higher scores indicate worse fatigue. Change score is computed by subtracting baseline Fatigue T-score from T-score at time of reassessment. Improvement is indicated by change scores with negative values.
Change in NIH Patient Reported Outcome Measures Information System (PROMIS) Fatigue, baseline to intermediate-term follow-up | Baseline collected between 3 months before start of stage 1 through 2 days after start of Stage 1. Intermediate-term follow-up measures collected between >6 month through <9 months after end of stage 2.
  PROMIS Fatigue reported in T-score, range 0-100, with 50 corresponding to the mean score and higher scores indicate worse fatigue. Change score is computed by subtracting baseline Fatigue T-score from T-score at time of reassessment. Improvement is indicated by change scores with negative values.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Flynn DM, McQuinn H, Fairchok A, Eaton LH, Langford DJ, Snow T, Doorenbos AZ. Enhancing the success of functional restoration using complementary and integrative therapies: Protocol and challenges of a comparative effectiveness study in active duty service members with chronic pain. Contemp Clin Trials Commun. 2018 Nov 29;13:100311. doi: 10.1016/j.conctc.2018.100311. eCollection 2019 Mar. PMID 30582069
- [Derived] Flynn DM, McQuinn H, Burke L, Steffen A, Fairchok A, Snow T, Doorenbos AZ. Use of Complementary and Integrative Health Therapies Before Intensive Functional Restoration in Active Duty Service Members with Chronic Pain. Pain Med. 2022 Apr 8;23(4):844-856. doi: 10.1093/pm/pnab326. PMID 34791423

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-07-09): https://cdn.clinicaltrials.gov/large-docs/40/NCT04656340/Prot_SAP_000.pdf
  • Informed Consent Form (2018-04-25): https://cdn.clinicaltrials.gov/large-docs/40/NCT04656340/ICF_001.pdf